CLINICAL TRIAL: NCT03932357
Title: Accuracy of Cone Beam Computed Tomography in Measuring of Mandibular Pig Soft Tissue Thickness Using a Radiopaque Material in Comparesion With Real Measurement.Diagnostic Study
Brief Title: Measuring Soft Tissue Thickness by CBCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahinaz Reda Hassan Abdelhamed, main supervisor Dr. Hoda Abd El Kader Saleh Professor, .Co-supervisor Dr: Walaa Abdelaty Associate Professor, Investigator: DR. Mahinaz Reda Hassan Assistant lecturer ., Cairo University
Other Study IDs: Mahinaz Reda
Record Dates: First submitted 2019-04-23; First posted 2019-04-30 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Cone Beam Computed Tomography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Radiation: CBCT — measuring soft tissue thickness using a CBCT

SUMMARY:
accuracy of CBCT in measuring soft tissue thickness by using a radiopaque material as the real finding and measurements on pig jaws

DETAILED DESCRIPTION:
* Pig jaws will be included in this study.
* Soft tissue surfaces were lightly covered with barium sulfate powder using a powder spray. CBCT was taken.
* A periodontal probe and a rubber stop were used for the measurement of trans-gingival probing thickness (TPT).
* After that, flap were elevated, and actual thickness of soft-tissue (actual thickness, AT) was measured.

The Analytical phase:

* In order to assess soft tissue thickness and bone levels an electronic digital caliper (Shenhan Measuring Tools Co., LTD, Shanghai) will used for measuring the transgingival probing thickness on the pig jaws.
* A graduated Naber's probe will be used for measuring the transgingival probing thickness.

Soft tissue thickness measurements:

* Intra-observer variability was tested under the supervision of the director.
* For the measurement of radiographic thickness (RT), wet soft tissue surfaces were covered with barium sulfate powder (SoloTop; Taejoon, Seoul, Korea), a radiopaque material used as a contrast medium.
* A probes and rubber stop were used for the measurement of transgingival probing thickness (TPT).
* A rubber stop was placed in contact with the surface to facilitate the measurement of tissue thickness, and then TPT was measured with digital calipers. All measurements were rounded to the nearest 0.01 mm.
* For the measurement of actual thickness (AT), an incision was made onto each marked area. After ﬂap elevation, actual soft tissue thickness was measured using the same method that was used for TPT.

Radiographic examination

* The pig jaws will then be imaged with CBCT.
* CBCT scanning will be performed using a PROMAX R 3DMid CBCT device (Planmeca Oy, Helsinki, Finland) with scanning protocol 90 kVp, 8 mA and 13.58 seconds exposure time with a single 360 degree rotation ROMEXIS software. The jawes will be placed on the horizontal plate of the device. The midline and mandibular position will be adjusted using the laser guide

ELIGIBILITY:
Inclusion Criteria:

* The study samples will not identified by age or gender group.
* The selected pig jaw should be intact with no mechanical damage.
* jaw with attached natural teeth

Exclusion Criteria:

* Teeth with anomalies and fractures.
* Periodontally affected teeth

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CBCT measuring soft tissue thickness using a radiopaque material
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2019-04-20 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-09 (Estimated)

PRIMARY OUTCOMES:
cbct | 6 months
  measuring soft tissue thickness using cbct in pig jaw

SECONDARY OUTCOMES:
Acutal thickness measurement | 6 months
  periodontal probe was inserted vertically into the soft tissue surface until resistance of the bone was felt
  . A rubber stop was placed in contact with the surface to facilitate the measurement of tissue thickness.actual thickness was measured with digital calipers

CONTACTS AND LOCATIONS:
Locations (1):
- Mahinaz Reda Hassan, Cairo, Giza-elharam, Egypt

IPD SHARING:
Plan to Share IPD: No